CLINICAL TRIAL: NCT01740713
Title: Multi-centre, Oral Single Dose Experimental and Modelling Study to Evaluate the Pharmacokinetics of Deferiprone in Patients Aged From 1 Month to Less Than 6 Years of Age Affected by Transfusion-dependent Haemoglobinopathies.
Brief Title: Pharmacokinetic Study of Deferiprone in Paediatric Patients
Acronym: DEEP-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Consorzio per Valutazioni Biologiche e Farmacologiche (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DEEP-1
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Iron Overload
Keywords: chronic iron overload; hereditary haemoglobinopathy; beta thalassaemia major
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferiprone; Isoflurophate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deferiprone, dose level 1 (Experimental): single dose level of 8.3 mg/kg every 8 hours for a corresponding total daily dose of 25 mg/kg/day.
  Interventions: Drug: Deferiprone, dose level 1
- Deferiprone, dose level 2 (Experimental): single dose level of 16.7 mg/kg every 8 hours for a corresponding total daily dose of 50 mg/kg/day.
  Interventions: Drug: Deferiprone, dose level 2
- Deferiprone, dose level 3 (Experimental): single dose level of 33.3 mg/kg every 8 hours for a corresponding total daily dose of 100 mg/kg/day.
  Interventions: Drug: Deferiprone, dose level 3

INTERVENTIONS:
Drug: Deferiprone, dose level 1 — a solution at 80 mg/mL will be administered orally
  Other Names: DFP
  Arms: Deferiprone, dose level 1
Drug: Deferiprone, dose level 2 — a solution at 80 mg/mL will be administered orally
  Other Names: DFP
  Arms: Deferiprone, dose level 2
Drug: Deferiprone, dose level 3 — a solution at 80 mg/mL will be administered orally
  Other Names: DFP
  Arms: Deferiprone, dose level 3

SUMMARY:
Deferiprone (DFP) is the most extensively studied oral iron chelator to date. It has been authorised in Europe in 1999 for the treatment of iron overload in patients with beta-thalassaemia major when DFO is contraindicated or inadequate. Despite a wide experience of DFP there are limited experimental data available on DFP in children and no pharmacokinetic data in children under 6 years of age. On the basis of the existing data in adults and adolescent, in the DEEP-1 trial a pharmacokinetic bridging model was developed to support the dose selection in children aged less than 6 years affected by transfusion dependent haemoglobinopathies. The study consisted of two phases, namely an experimental phase, during which patients received a single dose and a modeling phase, during which PK data obtained after single dose in patients < 6 years of age were analysed in conjunction with historical PK data in adults and older children and adolescents. The model-based analysis of the data obtained after single dose enabled the assessment of the dosing regimen required for the purpose of accurate pharmacokinetic bridging. The ratio between the predicted systemic exposure parameters (AUC and Cmax) in the target population and reference group were used as basis for recommendation of the dose in the target population.

DETAILED DESCRIPTION:
Deferiprone (DFP) was investigated as therapy for children from 1 month to less than 6 years of age. The study was a multicenter randomised, single blind, and single dose PK study. The patients were randomised according to a stratification scheme in which three different dose levels were used.

Objectives: The primary objective of this study was to assess the pharmacokinetics of DFP in paediatric patients aged from 1 month to less than 6 years.

The secondary objectives of this study were:

1. To identify dose levels yielding deferiprone exposures comparable to adults and define the dose rationale in children aged from 1 month to less than 6 years.
2. To evaluate safety and tolerability of deferiprone after single dose administration in children aged from 1 month to less than 6 years.
3. To evaluate the effect of demographic covariates on DFP disposition and estimate the clearance distribution across the population.

Endpoints: The primary endpoints of the study were pharmacokinetic and included:

* primary PK parameters: CL/F, Vd/F, Ka
* secondary PK parameters: AUC, Cmax, Tmax, Css and Cmin.

Secondary endpoints were assessment of clinical safety and tolerability .

Methods: Twenty-three patients were enrolled and 18 of those ( 9 males and 9 females) completed the study. The patients were administered at three dose levels ( 6 patients / each dose):

Dose level 1: 8.3 mg/kg as a single dose (every 8 h) for a total daily dose of 25mg/kg Dose level 2: 16.7 mg/kg as a single dose (every 8 h) for a total daily dose of 50 mg/kg Dose level 3: 33.3 mg/kg as a single dose (every 8 h) for a total daily dose of 100 mg/kg

Blood samples for PK analysis were taken at 6 sampling time intervals, different depending on the dose group: predose; in the range 10 -20 min; in the range 40-55min; in the range 1.05-1.15 h;in the range 1.25-5.30 h;in the range 6-8h after the first dose administration. The concentration of deferiprone was determined by a validated HPLC method. A population PK model approach was applied and the time course of deferiprone concentrations was analysed with Nonlinear mixed effects modelling in NONMEM, version 7.2.0. Model building included the assessment of the influence of relevant demographic covariates (i.e:body weight , age, height) on the disposition of deferiprone.

Using the pharmacokinetic model developed for the paediatric population in this study in conjunction with a model previously developed for 55 adult subjects , simulations were performed to evaluate drug exposure in children below 6 years of age and across a standard thalassaemic adult population.

Descriptive statistics were used to summarise adverse events, vital signs and clinical lab data (haematology, biochemistry and virology)

Results: A one-compartment model with first-order absorption was found to best describe the disposition of deferiprone. The choice of three dose levels enable to assess linearity of pharmacokinetic across the dose range. The disposition parameters estimated through the pop-PK model included CL/F , V/F. In addition to the final model parameter estimates, the secondary pharmacokinetic parameters were derived based on the individual predicted concentration vs. time profiles and were summarised per dose level.

Body weight was found to be a good predictor of inter-individual differences in the population under investigation.

As expected from the known safety profile of the drug, no Serious Adverse Events were observed during the DEEP-1 PK Study.

Based on the simulation analysis performed, a similar exposure is achieved in adults and children in terms of AUC and Css when receiving the current dosing regimen both at 75 and 100 mg/kg/day, while a considerable increase in Cmax was observed in children when compared to the adult population. However, exposure is the parameter related to clinical response rather than Cmax. Indeed, simulations suggested that a dosing regimen of 25 mg/kg t.i.d. (75 mg/kg/day) is recommended for children aged from 1 month to < 6 years, with the possibility of titration up to 33.3 mg/kg t.i.d. (100 mg/kg/day), if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients in a chronic transfusional program who have received at least 150 ml/kg/year of packed red blood cells (corresponding approximately to 12 transfusions) and on current treatment with DFO, DFX, DFP; aged from 1 month to less than 6 years; or
* Patients naïve to any chelation treatment who have received not less than 150 ml/kg of packed red blood cells (corresponding to approximately 12 transfusions) and have ferritin levels > 800 ng/mL, aged from 1 month to less than 6 years; or
* Patients who meet the transfusion criteria (150 ml/kg/year corresponding approximately to 12 transfusions) and have known intolerance or contraindication to DFO

And if all of the following criteria apply:

* Patients affected by any hereditary haemoglobinopathies requiring chronic transfusion therapy including but not limited to thalassaemia and sickle cell disease
* Written informed consent obtained from their legal guardian on the patient's behalf in accordance with the national legislations. According to his/her capability, patient's informed assent will be collected

Exclusion Criteria:

* Patient with known intolerance or contraindication to the trial treatment
* Patient with Hb levels less than 8g/dl (entry may be delayed until values return to normal)
* Patient with platelet count <100.000/mm3 or absolute neutrophil count <1.500/mm3 (entry may be delayed until values return to normal)
* Patient with evidence of abnormal liver function (ALT level >5 times the upper normal limit during six months preceding enrolment; entry may be delayed until values return to normal)
* iron overload from causes other than transfusional haemosiderosis
* severe heart dysfunction secondary to iron overload defined as the occurrence of heart failure or severe arrhythmia or as indicated by cardiac T2* lower than 10 ms, if recent MRI data is available,
* Patient with serum creatinine level above the upper normal limit at screening; entry may be delayed until values return to normal.
* Serological evidence of chronic hepatitis B (presence of HBe Ag, HBsAg, HBcAb-IgM, in the absence of HBsAb).
* History of significant medical or psychiatric disorder that may impair compliance with the requirements of the protocol.
* The patient has received another investigational drug within 30 days prior to this study.
* Patient with a pre-existing condition or any other surgical or medical condition which might significantly interfere with normal gastrointestinal and hepatic function that could alter the absorption, metabolism, and/or excretion of the study drug.
* Patient with a known history of HIV seropositivity.
* Fever and other signs/symptoms of infection in the 10 days before drug administration(treatment day)
* Concomitant use of other iron chelators or trivalent cation-dependent medicinal products such as aluminium-based antacids.
* Patient with a chronic condition that does not allow suspension of related treatment from starting of washout until drug is administered.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Della Pasqua, Study Chair — Universiteit Leiden, The Netherlands; Giovanni Carlo Del Vecchio, Principal Investigator — Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Italy
Locations (7):
- Department of Medical and Public Health Services of the Ministry of Health, Nicosia, Cyprus
- Cairo Univesity Paediatric Hospital, Cairo, Egypt
- Italy (5):
  - Azienda Ospedaliero-Universitaria Consorziale, Bari, Bari
  - Azienda Ospedaliera Antonio Cardarelli, Napoli, Napoli
  - Azienda Ospedaliera Di Padova, Padua, Padova
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo, Palermo
  - Clinica Pediatrica Universita' - Asl 1, Sassari, Sassari

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 children affected by transfusion-dependent haemoglobinopathies were enrolled in this study. Of these 23 children, 2 were screening failures and 3 early terminations.
Groups:
- Deferiprone 25 mg/kg/Day: Deferiprone will be administered at 25 mg/kg/day
  Deferiprone, dose level 1: deferiprone liquid oral solution (80 mg/ml)
- Deferiprone 50 mg/kg/da: Deferiprone will be administered at 50 mg/kg/day
  Deferiprone, dose level 2: deferiprone liquid oral solution (80 mg/ml)
- Deferiprone 100 mg/kg/Day: Deferiprone will be administered at 100 mg/kg/day
  Deferiprone, dose level 3: deferiprone liquid oral solution (80 mg/ml)
Period: Overall Study
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/da | Deferiprone 100 mg/kg/Day
Started | 6 | 8 | 7
Completed | 6 | 6 | 6
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Deferiprone 50 mg/kg/Day: Deferiprone will be administered at 50 mg/kg/day
  Deferiprone, dose level 2: deferiprone liquid oral solution (80 mg/ml)
- Total: Total of all reporting groups
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day | Total
Number analyzed (Participants) | 6 | 8 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 8 | 7 | 21
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 3 | 4 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Italy | 6 | 8 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: CL/F
Description: Plasma clearance after oral administration. The parameter was estimated through a population pharmacokinetic model, during which concentration data obtained after single oral dose ( at 3 dose levels) of DFP in patients aged from 1 month to less than 6 years of age.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Mean (Standard Error); unit: litre/h
Groups:
- PK Population: Deferiprone liquid oral solution (80 mg/ml) has been administered at 25/50/100 mg/kg/day
Arm/Group | PK Population
Number analyzed (Participants) | 18
litre/h | 8.3 (0.569)

2. Primary Outcome: AUC (0-8h)
Description: Area under concentration versus time curve from 0 to 8 h post dosing. Secondary pharmacokinetic parameter derived on the basis of the individual predicted concentration vs. time profiles, through the pop-PK model.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Median (Inter-Quartile Range); unit: micromol*h/L
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day
Number analyzed (Participants) | 6 | 6 | 6
micromol*h/L | 116.7 [90.6 to 129.0] | 210.0 [173.1 to 266.6] | 428.8 [291.4 to 547.8]

3. Primary Outcome: V/F
Description: volume of distribution after oral administration. The parameter was estimated through a population pharmacokinetic model, during which concentration data obtained after single oral dose ( at 3 dose levels) of DFP in patients aged from 1 month to less than 6 years of age
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Mean (Standard Error); unit: litres
Arm/Group | PK Population
Number analyzed (Participants) | 18
litres | 18.7 (1.16)

4. Primary Outcome: Tmax
Description: Time at which the maximum concentration (Cmax) is reached. Secondary pharmacokinetic parameters such as Cmax, Min, Tmax, Css and AUC (0-8h) were derived based on the individual predicted concentration vs. time profiles.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day
Number analyzed (Participants) | 6 | 6 | 6
hour | 0.33 [0.19 to 0.92] | 0.33 [0.21 to 0.63] | 0.37 [0.27 to 0.42]

5. Primary Outcome: Ka
Description: Absorption rate constant. The parameter was estimated through a population pharmacokinetic model, during which concentration data obtained after single oral dose ( at 3 dose levels) of DFP in patients aged from 1 month to less than 6 years of age.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Mean (Standard Error); unit: h^-1
Arm/Group | PK Population
Number analyzed (Participants) | 18
h^-1 | 9.13 (1.41)

6. Primary Outcome: Cmax
Description: Maximum concentration reached in plasma. Secondary pharmacokinetic parameter derived on the basis of the individual predicted concentration vs. time profiles, through the pop-PK model.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Median (Inter-Quartile Range); unit: microM
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day
Number analyzed (Participants) | 6 | 6 | 6
microM | 61.7 [45.1 to 80.7] | 119.8 [106 to 154] | 229.5 [179.7 to 278.1]

7. Primary Outcome: Css
Description: Plasma concentration reached at steady state. Secondary pharmacokinetic parameter derived on the basis of the individual predicted concentration vs. time profiles, through the pop-PK model.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Median (Inter-Quartile Range); unit: microM
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day
Number analyzed (Participants) | 6 | 6 | 6
microM | 2.1 [1.6 to 2.3] | 3.7 [3.1 to 4.9] | 7.7 [5.1 to 10]

8. Primary Outcome: Cmin
Description: Minimum plasma concentration. Secondary pharmacokinetic parameter derived on the basis of the individual predicted concentration vs. time profiles, through the pop-PK model.
Time Frame: Day 1 of single dose treatment (6 sampling time range: from predose up to 8h post first administration)
Measure: Median (Inter-Quartile Range); unit: microM
Arm/Group | Deferiprone 25 mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day
Number analyzed (Participants) | 6 | 6 | 6
microM | 1.5 [0.92 to 2.6] | 1.9 [0.79 to 5.5] | 6.8 [3.1 to 13.9]

9. Secondary Outcome: Adverse Events
Description: All the medical occurrences that started after the administration of the drug
Time Frame: from drug administration up to 8 days post treatment
Measure: Number; unit: participants
Groups:
- Safety Population: patients who may experience adverse events occurred before or after treatment
Arm/Group | Safety Population
Number analyzed (Participants) | 21
participants | 3

ADVERSE EVENTS:
Time Frame: All the medical occurrences that started after the administration of the drug under investigation have been recorded as AEs till the follow -up visit at 8 days post dosing.
Groups:
- Deferiprone 25mg/kg/Day: Deferiprone will be administered at 25 mg/kg/day
  Deferiprone, dose level 1: deferiprone liquid oral solution (80 mg/ml)
Arm/Group | Deferiprone 25mg/kg/Day | Deferiprone 50 mg/kg/Day | Deferiprone 100 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/6 | 0/8 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone 25mg/kg/Day (N=6) | Deferiprone 50 mg/kg/Day (N=8) | Deferiprone 100 mg/kg/Day (N=7)
Infantile spitting up (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Rash trunk (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No